CLINICAL TRIAL: NCT07142174
Title: Improving Cervical Spine Alignment and Intervertebral Foramen Expansion Using a Novel Distally Expanding Cervical Facet Implant (CeLFI) for Cervical Degenerative Disease
Brief Title: Improving Cervical Spine Alignment and Intervertebral Foramen Expansion Using a Novel Distally Expanding Cervical Facet Implant for Cervical Degenerative Disease
Acronym: CeLFI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Amro Fayez Alhabib, Professor of Neurosurgery, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-21-6224; 2329 (Other: Saudi FDA)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cervical Degenerative Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible Patients (Experimental): Patients who met the inclusion criteria and will go to intervention.
  Interventions: Device: cervical facet implant will be introduced into the cervical levels that were mobile on flexion-extension x-ray and exhibited foramen stenosis or spondylolisthesis

INTERVENTIONS:
Device: cervical facet implant will be introduced into the cervical levels that were mobile on flexion-extension x-ray and exhibited foramen stenosis or spondylolisthesis — The patients will be managed according to the current practice for posterior cervical spine surgical approaches regarding patient positioning, surgical exposure, and neural decompression. The patients will be positioned prone with the head in a Mayfield headrest, All patients will be monitored using intraoperative motor evoked potentials (MEP) and somatosensory evoked potentials (SSEP). Intra-operative X-rays (antero-posterior and lateral) will be used to identify the index cervical level and to guide facet preparation and CeLFI insertion. Exposure of the posterior surface of the lateral mass at the index level of the cervical spine will be done either through a midline open technique or para-midline; inter-muscular approach (MIS). The facet joint-space (FJS) will be opened using a monopolar cautery with careful attention to preserve the joint's capsule on the lateral and medial boundaries.
  The FJS will be prepared using sequential dilators; designed for this purpose. Each dilator me

SUMMARY:
Cervical degenerative disease (CDD) resulting in myelopathy represents the commonest disease affecting the spinal cord in adults. Cervical radiculopathy can be associated with myelopathy or occurs alone. The treatment frequently requires surgical intervention; which could be done through anterior or posterior cervical spine approach, or a combination. In this study, we aim to evaluate the value of the innovative device (CeLFI; Cervical expanding facet implant), inserted from posterior approach, in widening the neural intervertebral foramina by providing an anterior distraction of the cervical facet joint space (FJS). Therefore, achieving indirect nerve decompression while maintaining cervical alignment and stability.

A prospective clinical study of a biomechanically and cadaver-validated device, following the pathway of similarly approved devices. Informed consent will be taken before the participation of every patient. 20 adult patients undergoing posterior surgery for CDD (for radiculopathy or myelopathy); from C2-6, will be included. Clinical evaluation will include pre- and post-operative standard outcome measures including visual analogue score (VAS), Neck disability index (NDI), and Modified Japanese Orthopedic Association score (mJOA). Standard radiologic evaluation will be performed before and after surgery including X-ray, computer tomography scan (CT), and Magnetic resonance imaging (MRI). Interim detailed safety analysis will be conducted after the first 5 cases are performed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Signed Informed Consent
* Patients undergoing posterior cervical Spine surgery for CDD (for radiculopathy or myelopathy)

Exclusion Criteria:

* Non-degenerative cervical spine pathologies, including infection, tumor, or trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
• Primary outcome (Radiological Evaluation): o Reduction of spondylolisthesis segment on X-rays (both intra-operative and post-operative within 1 week from surgery). This is defined here as a reduction of prior cervical vertebral mal-alignment to less t | 1, 3, and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No